CLINICAL TRIAL: NCT04854473
Title: Data Collection Study - Recording Electro-physiological Signals From Intact (to be Resected, Pathological) and Ischemic Bowel Tissue During Open Colonic Surgery.
Brief Title: Collection of Electrophysiological Data During Colon Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exero Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLP-01
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Open/ Laparoscopic/ Robotic Resection of the Colon
Keywords: Exero; anastomotic leak; impedance; ischemia; colon; bowel
MeSH Terms: conditions — Anastomotic Leak; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance measurement (Experimental): Subjects with Exero's Smart Drain Device Attached This arm contains subjects which will have Exero's leak detection Device used: Exero Smart Drain is placed on their large bowel during colonic resection surgery (either open, laparoscopic or robotic). The study aims to demonstrate that the parameters measured by the device in in-vivo, non-disrupted tissue are different than parameters measured in ischemic tissue. Once this data is collected a detection algorithm can be trained. This procedure will add no more than 20 minutes to the existing procedure that is performed per hospital standard overall and will enable collection of control vs. ischemia induced clinical data, essential to developing the detection algorithms.
  Interventions: Device: Exero Medical Leak Detection System

INTERVENTIONS:
Device: Exero Medical Leak Detection System — the Exero Leak Detection System components used in this study are:
  * Smart drain - a surgical drain with added sensing electrodes
  * Transceiver /Recording Unit (TRU) - a wearable placed outside the body on intact skin and is connected to the implanted electrodes. The unit also acts as a wireless connection to the Monitoring Subsystem.
  * Monitoring Subsystem - a tablet or a computer connected wirelessly to the transceiver providing logging, applying analysis algorithms on the logged signals and providing indication/alerts to the medical staff derived from the signals recorded by the electrodes.

SUMMARY:
The study is conducted to record continuous electrophysiological signals from intact and ischemic bowel tissue during colonic resection surgery, in order to train the Exero Medical Leak Detection System classification algorithm on detection of ischemic conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient is scheduled for open colonic resection, (right hemicolectomy, left hemicolectomy, sigmoidectomy, anterior resection or subtotal colectomy) surgery.
3. Patient has consented to be in the trial and signed informed consent is available before any study related procedures are carried out.

Exclusion Criteria:

1. Subject has gastroparesis.
2. Subject has significant multisystem (autonomic) diseases.
3. Subject has a body mass Index greater than 35 kg/m2
4. Subject has an autoimmune disorder requiring therapy in the preceding 2 years.
5. Subject has significant cardiac arrhythmia or ectopy.
6. Obstructing lesion and pre obstruction bowel dilatation
7. Subject has an existing implanted electrical stimulator (e.g., pacemaker.
8. Subject requires chronic anticoagulant therapy
9. Subject is currently enrolled in other potentially confounding research.
10. Pregnancy
11. Current alcohol abuse
12. Subject poses a significant general anesthesia risk
13. Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Functionality of signal measurement | 10 minutes
  Baseline data collected from the intended bowel segment to be resected, prior to tissue manipulation, is compared to the data recorded after the ischemia induced by the resection procedure.

SECONDARY OUTCOMES:
Occurrence of adverse events | 10 minutes
  Adverse events both expected and unexpected, related or unrelated to study device or procedure, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Nir Wasserberg, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No